CLINICAL TRIAL: NCT00005372
Title: Intimal Thickening and Antioxidants in Hispanics and Anglos (Los Angeles Atherosclerosis Study)
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4264; R01HL049910 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To investigate the role of serum and dietary antioxidants, serum pro-oxidants, and smoking on the progression/regression of carotid intima-media thickness (IMT).

DETAILED DESCRIPTION:
BACKGROUND:

A finding from the Cholesterol Lowering Atherosclerosis Study (CLAS), a clinical trial, indicated that common carotid intima-media thickness responded more rapidly and more markedly to LDL-C lowering treatment than angiographic coronary stenosis or carotid roughness. New data from a primate model also showed ultrasound detection of intimal thickening in response to a hypercholesterolemic diet within twelve months. These findings suggest that carotid IMT is a reliable and rapidly responding marker of extent of atherosclerosis. However, less than a third of the observed therapeutic benefit on carotid IMT found in CLAS was explained by change in LDL-C and HDL-C, suggesting that related (or other) factors are more directly linked to atherogenic mechanisms. In addition, a Finnish epidemiologic study found that LDL-C was predicative of rate of progression in carotid IMT only in persons with high serum levels of (pro-oxidant) copper. . These and other data support a model of atherosclerosis in which intracellular accumulation of modified LDL is promoted/retarded by serum pro-oxidants/antioxidants.

DESIGN NARRATIVE:

The study tested the specific hypotheses that the positive association between rate of increase in carotid IMT and low density lipoprotein cholesterol (beta deltaIMT/LDL) was greater in persons with [1] higher levels of serum pro-oxidants (relative to persons with lower levels of serum pro-oxidants), [2] lower levels of serum antioxidants, [3] lower levels of dietary antioxidants; and [4] that regression of carotid IMT associated with smoking cessation would be detected in 30 months. Hypothesis were tested with the longitudinal observation of carotid IMT in Hispanic and non-Hispanic white women and men. The inclusion of Hispanics and women was motivated by their prevalence in the study population (18 percent Hispanic, 40 percent women), and by the then recent report that incidence of hospitalization for myocardial infarction was elevated in Hispanics. Seventy three persons from each of four ethnicity-sex groups aged 40-60 years (n-292), and 83 smokers and recent quitters (n-166) were recruited from employees in an ongoing study. Baseline blood, diet and potential confounder variables were related to 18 and 36 month (6, 12, 18, 24 and 30 month in smoker(s) changes in carotid IMT. Levels of antioxidant vitamins, including alpha-tocopherol, ascorbate, and beta carotene, in the plasma were measured at baseline. Plasma levels of negatively charged LDL were measured in a sub-sample of subjects with the most rapidly progressing common carotid intima-media thickness and in an age-sex matched subsample with the least rapidly progressing common carotid intima-media thickness. Finally, an ultrasound measurement of carotid arterial stiffness, another indicator of early atherosclerosis, was developed to address the role of blood pressure.

The Los Angeles Atherosclerosis Study (LAAS) has been renewed through February, 2004 to continue follow-up of the cohort for a total of seven years with two additional measures of arterial dysfunction, including endothelial function of the brachial artery and distensibility or stiffness of the common carotid artery.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-01; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: James Dwyer — University of Southern California

REFERENCES:
- [Background] Dwyer JH. Exposure to environmental tobacco smoke and coronary risk. Circulation. 1997 Sep 2;96(5):1367-9. No abstract available. PMID 9315516
- [Background] Dwyer JH, Sun P, Kwong-Fu H, Dwyer KM, Selzer RH. Automated intima-media thickness: the Los Angeles Atherosclerosis Study. Ultrasound Med Biol. 1998 Sep;24(7):981-7. doi: 10.1016/s0301-5629(98)00069-6. PMID 9809632
- [Background] Nordstrom CK, Dwyer KM, Merz CN, Shircore A, Dwyer JH. Work-related stress and early atherosclerosis. Epidemiology. 2001 Mar;12(2):180-5. doi: 10.1097/00001648-200103000-00009. PMID 11246578
- [Background] Sun P, Dwyer KM, Merz CN, Sun W, Johnson CA, Shircore AM, Dwyer JH. Blood pressure, LDL cholesterol, and intima-media thickness: a test of the "response to injury" hypothesis of atherosclerosis. Arterioscler Thromb Vasc Biol. 2000 Aug;20(8):2005-10. doi: 10.1161/01.atv.20.8.2005. PMID 10938024
- [Background] Dwyer KM, Nordstrom CK, Bairey Merz CN, Dwyer JH. Carotid wall thickness and years since bilateral oophorectomy: the Los Angeles Atherosclerosis Study. Am J Epidemiol. 2002 Sep 1;156(5):438-44. doi: 10.1093/aje/kwf051. PMID 12196313
- [Background] Bairey Merz CN, Dwyer J, Nordstrom CK, Walton KG, Salerno JW, Schneider RH. Psychosocial stress and cardiovascular disease: pathophysiological links. Behav Med. 2002 Winter;27(4):141-7. doi: 10.1080/08964280209596039. PMID 12165968
- [Background] Nordstrom CK, Dwyer KM, Merz CN, Shircore A, Dwyer JH. Leisure time physical activity and early atherosclerosis: the Los Angeles Atherosclerosis Study. Am J Med. 2003 Jul;115(1):19-25. doi: 10.1016/s0002-9343(03)00242-0. PMID 12867230
- [Background] Dwyer JH, Navab M, Dwyer KM, Hassan K, Sun P, Shircore A, Hama-Levy S, Hough G, Wang X, Drake T, Merz CN, Fogelman AM. Oxygenated carotenoid lutein and progression of early atherosclerosis: the Los Angeles atherosclerosis study. Circulation. 2001 Jun 19;103(24):2922-7. doi: 10.1161/01.cir.103.24.2922. PMID 11413081
- [Background] Dwyer JH, Allayee H, Dwyer KM, Fan J, Wu H, Mar R, Lusis AJ, Mehrabian M. Arachidonate 5-lipoxygenase promoter genotype, dietary arachidonic acid, and atherosclerosis. N Engl J Med. 2004 Jan 1;350(1):29-37. doi: 10.1056/NEJMoa025079. PMID 14702425
- [Background] Wu H, Dwyer KM, Fan Z, Shircore A, Fan J, Dwyer JH. Dietary fiber and progression of atherosclerosis: the Los Angeles Atherosclerosis Study. Am J Clin Nutr. 2003 Dec;78(6):1085-91. doi: 10.1093/ajcn/78.6.1085. PMID 14668268
- [Background] Burcelin R, Eddouks M, Kande J, Assan R, Girard J. Evidence that GLUT-2 mRNA and protein concentrations are decreased by hyperinsulinaemia and increased by hyperglycaemia in liver of diabetic rats. Biochem J. 1992 Dec 1;288 ( Pt 2)(Pt 2):675-9. doi: 10.1042/bj2880675. PMID 1463468